CLINICAL TRIAL: NCT00157651
Title: A Double-Blind, Placebo Controlled, Randomized Trial of Low-Intensity Adjusted-Dose Warfarin for the Prevention of Mechanical Malfunction of Double-Lumen Haemodialysis Catheters
Brief Title: Access II - Trial of Warfarin to Prevent Malfunction of Haemodialysis Catheters
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Dr. Alistair Ingram Professor of Medicine, McMaster University
Organization: McMaster University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MCT-15226
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2008-06-17 (Estimated); Status verified 2008-06

CONDITIONS: End Stage Renal Disease; Thrombosis; Bleeding
Keywords: end stage renal disease; thrombosis; bleeding
MeSH Terms: conditions — Kidney Failure, Chronic; Thrombosis; Hemorrhage | interventions — Warfarin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Receiving warfarin
  Interventions: Drug: warfarin
- 2 (Placebo Comparator): Receiving matching placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: warfarin — Daily oral warfarin with INR monitored weekly, adjusted to keep INR between 1.5 and 1.9
  Other Names: Coumadin
  Arms: 1
Drug: placebo — matching placebo for warfarin, adjusted according to sham INR generated by unblinded warfarin monitor
  Other Names: no other names
  Arms: 2

SUMMARY:
This study examines whether low intensity, dose adjusted warfarin prolongs the time to mechanical failure of hemodialysis catheters without resulting in an unacceptable rate of bleeding.

DETAILED DESCRIPTION:
Patients with end-stage renal disease receiving or about to initiate hemodialysis are randomized to receive either adjusted dose warfarin to achieve an INR of 1.5-1.9 or adjusted dose placebo within 72 hours of hemodialysis catheter placement. The primary outcome is mechanical failure of the catheter, as outlined below.

ELIGIBILITY:
Inclusion Criteria:

* Newly placed double-lumen hemodialysis catheter

Exclusion Criteria:

* Major bleed within last 3 months
* Platelet count less than 50 x 10 9/L or current coagulopathy (most recent INR > 1.5, not due to warfarin)
* Active peptic ulcer disease
* Anticipated need for invasive intervention within next 2 weeks
* Taking warfarin for an indication other than access prophylaxis
* Allergic to, or intolerant of, warfarin
* Pregnant
* Woman of child-bearing age who has not agreed to use an adequate method of birth control for the duration of the study
* Catheter likely needed for 2 weeks or less
* Patient previously took part in the study
* Patient has known aortic aneurysm of 6cm or greater
* Patients nephrologist has refused consent
* Patient has refused consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 1999-02; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Time from catheter insertion to mechanical failure. This is defined as inability to aspirate or persistent blood flow less than 200mL/min after line reversal, patient repositioning and rotational manipulation of the catheter. | monthly

SECONDARY OUTCOMES:
Blood flow rate and adequacy of dialysis. | monthly
Major bleeding events. | monthly
Death from any cause. | monthly

CONTACTS AND LOCATIONS:
Overall Officials: Alistair J Ingram, MD, Principal Investigator — Associate Professor, Medicine; Catherine M Clase, MD, Principal Investigator — Associate Professor, Medicine
Locations (1):
- St. Joseph's Healthcare, Hamilton, Ontario, Canada